CLINICAL TRIAL: NCT06966427
Title: Prospective Evaluation of a Dose Guidance System for People With Diabetes Initiating Basal Insulin or Using Insulin Injections
Acronym: DGS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: DreaMed Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0023-25-RMC
Record Dates: First submitted 2025-04-29; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Type 1 diabetes; Type 2 diabetes; Dose guidance system
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, single blind, two-arms, multicenter study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dosing Guidance System- Group A (Experimental): Any insulin dosing event manually logged by the participant, the DGS will receive the time and amount of the dose as input.
  Interventions: Device: Dosing Guidance System to be used with both time and amount of insulin as input
- Dosing Guidance System-Group B (Experimental): Any insulin dosing event manually logged by the participant, the DGS will receive only the time of the dose as input
  Interventions: Device: Dosing Guidance System to be used with only time of insulin as input

INTERVENTIONS:
Device: Dosing Guidance System to be used with both time and amount of insulin as input — Any insulin dosing event manually logged by the participant, the DGS will receive the time and amount of the dose as input
  Other Names: endo.digital (Modi algorithm)
  Arms: Dosing Guidance System- Group A
Device: Dosing Guidance System to be used with only time of insulin as input — any insulin dosing event manually logged by the participant, the DGS will receive only the time of the dose as input
  Other Names: endo.digital (Modi algorithm)
  Arms: Dosing Guidance System-Group B

SUMMARY:
A prospective, randomized, single blind, two-arms, multicenter study. The study aims to assess the safety of a dosing-guided system (DGS) that provides direct advice on insulin dosing recommendations and diabetes management to individuals with diabetes using insulin or starting basal insulin therapy, guided by their continuous glucose monitoring (CGM).

The study population will include up to 45 individuals with diabetes, distributed as follows: 15 with Type 1 diabetes (T1D) and 15 with Type 2 diabetes (T2D), both on MDI therapy and 15 with T2D using or starting to use basal insulin.

The study will include a 2- to 4-week run-in period followed by a 6-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Documented T1D or T2D, for at least 6 months
* Aged ≥ 6 years ≤ 75 years
* HbA1c ≤ 11%
* For Segment 1: Using basal-bolus MDI therapy, i.e. basal insulin and a bolus that is either:

  1. Carbohydrate counting with carbohydrate ratio (CR) and correction factor (CF)
  2. Fix dose for meal / meal estimation with CF
* For Segment 2: Using or prescribed basal insulin
* Participants using the following type of insulin as directed in the instructions for use:

  1. Basal insulin: Glargine (including Rezvoglar, Semglee, Toujeo, Soliqua), Degludec (including Tresiba U-100, Tresiba U-200, Xultophy), Determir
  2. Bolus insulin: regular insulin, rapid analogues (Insulin Aspart, Insulin Glulisine, Insulin Lispro) or ultra-rapid analogues (Fiasp, Lyumjev)
* Participants willing to use FreesStyle Libre CGM according to manufacturer instructions, document insulin delivery, meals, and daily activities.
* Participants have a smartphone compatible with study requirements.
* Participants are willing and able to sign a written informed consent form to use their data.
* Participants are willing to use the bolus calculator for insulin dosing (only for segment 1)

Exclusion Criteria:

1. Concomitant diseases/treatment that influence metabolic control or any significant diseases/conditions including psychiatric disorders and substance abuse or drug or alcohol abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patients' safety.
2. Relevant severe organ disorders (diabetic nephropathy, diabetic retinopathy, diabetic foot syndrome) or any secondary disease or complication of diabetes mellitus, such as:

   1. Subject has unstable or rapidly progressive renal disease or has eGFR < 45 or is receiving dialysis
   2. Subject has active proliferative retinopathy
   3. Active gastroparesis
3. Participation in any other interventional study
4. Female participant who is pregnant or planning to become pregnant within the planned study duration
5. Individuals who are using one of the following types of insulin:

   1. Intermediate-acting insulin (NPH)
   2. Mixed insulin like:

   i. Premix NPH/ Regular (e.g. Humalin 70/30, Novolog 70/30) ii. Premix analogs (e.g, Novolog mix 70/30, Hu,alog mix 75, 25, Humalog Mix 50/50) c. Inhale insulin (e.g. Afrezza)
6. Hypoglycemia unawareness
7. Individuals who are treated with intravenous (IV) insulin injections, or a combination of insulin injections and/or IV insulin and insulin pump therapy.
8. Individuals who have extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements.
9. An episode of diabetic keto-acidosis within the month prior to study entry and/or severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrolment.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Sensor glucose percentage of time in hypoglycemia below 54 mg/dL | Aafter 6 weeks of intervention period
  Will be compared between the last two weeks of the run-in period and the last two weeks of the intervention

SECONDARY OUTCOMES:
Number of events of glucose readings below 54 mg/dL | After 6 weeks of intervention period
  An event is defined as a period of at least 15 minutes of glucose readings below 54 mg/dL.
  Will be compared between the last two weeks of the run-in period and the last two weeks of the intervention
Sensor glucose percentage of time in hyperglycemia above 250 mg/dL | After 6 weeks of intervention period
  Will be compared between the last two weeks of the run-in period and the last two weeks of the intervention

OTHER OUTCOMES:
Glucose Management Indicator (GMI) | After 6 weeks of intervention period
Percentage of glucose readings between 70- 180 mg/dl | After 6 weeks of intervention period
  Will be compared between the last two weeks of the run-in period and the last two weeks of the intervention
Change in (Hemoglobin A1c) HbA1C post-study treatment | After 6 weeks of intervention period
Percentage of glucose readings below 70 mg/dl | After 6 weeks of intervention period
  Will be compared between the last two weeks of the run-in period and the last two weeks of the intervention
Mean sensor glucose | After 6 weeks of intervention period
  Will be compared between the last two weeks of the run-in period and the last two weeks of the intervention
Glucose variability measured by Standard Deviation (SD) and CV% | After 6 weeks of intervention period
  Will be compared between the last two weeks of the run-in period and the last two weeks of the intervention
Time to reach optimal insulin dose | After 6 weeks of intervention period
Total insulin dose and the amount of basal and/or bolus insulin dose | After 6 weeks of intervention period
Device satisfaction questioner | After 6 weeks of intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, MD, Principal Investigator — Schneider Children's Medical Center
Locations (2):
- Schneider Children Medical Center of Israel, Petah Tikva, Israel
- University Medical Center of Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No